CLINICAL TRIAL: NCT04250441
Title: The Use of Transcranial Focused Ultrasound for the Treatment of Depression and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32222-2
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): All patients enrolled will receive transcranial focused ultrasound. Target location is dependent on patient condition.
  Interventions: Device: Focused Transcranial Ultrasound

INTERVENTIONS:
Device: Focused Transcranial Ultrasound — The FDA has determined that power intensity limits of 720 mW/cm squared at 2 megaHertz is safe for clinical use; the proposed equipment works within these parameters. Furthermore, monitoring sessions up to one hour as proposed in this study are routinely used in patients even with acute brain injury at 2 megaHertz without any reports of complications induced by the ultrasound device. No brain heating, cavitation or bleeding has been identified with the proposed equipment and protocol. For each individual safety can be followed by performing a selective mental status exam at each session completion.

SUMMARY:
The purpose of this open label study is to evaluate longer term tolerability and early efficacy of transcranial ultrasound in the treatment of patients with refractory depression and anxiety.

DETAILED DESCRIPTION:
The present study is designed as an open label study of patients with refractory depression and anxiety to evaluate longer term tolerability and early efficacy of transcranial ultrasound treatment. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures which are not affected by practice effects. For patients with refractory depression, the target will be the subgenual cingulate (Brodmann's area 25) through a trans temporal scalp window. For patients with anxiety, the target will be the amygdala. Targeting will include reference to scalp fiducials based on the obtained MRI and Doppler waveform confirmation will be obtained because of the ability of TCD to record Doppler signal from the posterior cerebral artery that runs medial to the mesial temporal lobe.

On the day of the ultrasound appointment, patients will undergo ten to thirty minutes of transcranial ultrasound treatment. The sonification device will be aimed at the subgenual cingulate or amygdala, depending on the predetermined condition. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space. Patients will undergo 8 total sessions of focused ultrasound. Patients will be evaluated at baseline and upon final ultrasound treatment using the same measures obtained upon entry. Safety and any adverse events will be monitored closely.

ELIGIBILITY:
Inclusion Criteria for Depression:

* Diagnosis of Major Depressive Disorder
* Score greater than 13 on the Beck Depression Inventory
* Failure to remit with 3 antidepressants
* At least 18 years of age

Inclusion Criteria for Anxiety:

* Diagnosis of Generalized or Acute Anxiety Disorder
* Score greater than 15 on the Beck Anxiety Inventory
* Failure to remit with 3 anxiolytics
* At least 18 years of age

Exclusion Criteria for Depression & Anxiety:

* Cognitive decline clearly related to an acute illness
* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Recent surgery or dental work within 3 months of the scheduled procedure.
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Any active cancer or chemotherapy
* Any other neoplastic illness or illness characterized by neovascularity
* Macular degeneration
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced kidney, pulmonary, cardiac or liver failure

Ages: 18 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline prior to ultrasound administration (
  [Primary for patients enrolled for depression] The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Hamilton Anxiety Rating Scale | Baseline prior to ultrasound administration
  [Primary for patients enrolled for anxiety] The HAM-A is an observer/rater scale consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | After final ultrasound (8 weeks from baseline)
  [Administered to patients enrolled with anxiety] The HAM-A is an observer/rater scale consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Beck Anxiety Inventory | Baseline prior to ultrasound administration
  [Administered to patients enrolled with anxiety] The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Anxiety Inventory | After final ultrasound (8 weeks from baseline)
  [Administered to patients enrolled with anxiety] The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Patient Depression Questionnaire | After final ultrasound (8 weeks from baseline)
  [Administered to patients enrolled with depression] The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
Hamilton Depression Rating Scale | Baseline prior to ultrasound administration
  [Administered to patients enrolled with depression] The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
Hamilton Depression Rating Scale | After final ultrasound (8 weeks from baseline)
  [Administered to patients enrolled with depression] The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
Beck Depression Inventory | After final ultrasound (8 weeks from baseline)
  [Administered to patients enrolled with depression] The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, M.D., Principal Investigator — Neurological Associates - the Interventional Group
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Background] Montgomery SA, Baldwin DS, Riley A. Antidepressant medications: a review of the evidence for drug-induced sexual dysfunction. J Affect Disord. 2002 May;69(1-3):119-40. doi: 10.1016/s0165-0327(01)00313-5. PMID 12103459
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Cipriani A, Furukawa TA, Salanti G, Geddes JR, Higgins JP, Churchill R, Watanabe N, Nakagawa A, Omori IM, McGuire H, Tansella M, Barbui C. Comparative efficacy and acceptability of 12 new-generation antidepressants: a multiple-treatments meta-analysis. Lancet. 2009 Feb 28;373(9665):746-58. doi: 10.1016/S0140-6736(09)60046-5. PMID 19185342
- [Background] Setiawan E, Attwells S, Wilson AA, Mizrahi R, Rusjan PM, Miler L, Xu C, Sharma S, Kish S, Houle S, Meyer JH. Association of translocator protein total distribution volume with duration of untreated major depressive disorder: a cross-sectional study. Lancet Psychiatry. 2018 Apr;5(4):339-347. doi: 10.1016/S2215-0366(18)30048-8. Epub 2018 Feb 26. PMID 29496589
- [Background] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Background] Lozano AM, Mayberg HS, Giacobbe P, Hamani C, Craddock RC, Kennedy SH. Subcallosal cingulate gyrus deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):461-7. doi: 10.1016/j.biopsych.2008.05.034. Epub 2008 Jul 18. PMID 18639234
- [Background] Jalbrzikowski M, Larsen B, Hallquist MN, Foran W, Calabro F, Luna B. Development of White Matter Microstructure and Intrinsic Functional Connectivity Between the Amygdala and Ventromedial Prefrontal Cortex: Associations With Anxiety and Depression. Biol Psychiatry. 2017 Oct 1;82(7):511-521. doi: 10.1016/j.biopsych.2017.01.008. Epub 2017 Jan 17. PMID 28274468
- [Background] Mayberg H. Depression, II: localization of pathophysiology. Am J Psychiatry. 2002 Dec;159(12):1979. doi: 10.1176/appi.ajp.159.12.1979. No abstract available. PMID 12450943
- [Background] Mayberg HS. Limbic-cortical dysregulation: a proposed model of depression. J Neuropsychiatry Clin Neurosci. 1997 Summer;9(3):471-81. doi: 10.1176/jnp.9.3.471. PMID 9276848
- [Background] Mayberg HS. Modulating limbic-cortical circuits in depression: targets of antidepressant treatments. Semin Clin Neuropsychiatry. 2002 Oct;7(4):255-68. doi: 10.1053/scnp.2002.35223. PMID 12382208
- [Background] Mayberg HS. Modulating dysfunctional limbic-cortical circuits in depression: towards development of brain-based algorithms for diagnosis and optimised treatment. Br Med Bull. 2003;65:193-207. doi: 10.1093/bmb/65.1.193. PMID 12697626
- [Background] Mayberg HS. Positron emission tomography imaging in depression: a neural systems perspective. Neuroimaging Clin N Am. 2003 Nov;13(4):805-15. doi: 10.1016/s1052-5149(03)00104-7. PMID 15024963
- [Background] Mayberg HS. Defining the neural circuitry of depression: toward a new nosology with therapeutic implications. Biol Psychiatry. 2007 Mar 15;61(6):729-30. doi: 10.1016/j.biopsych.2007.01.013. No abstract available. PMID 17338903
- [Background] Mayberg HS. Targeted electrode-based modulation of neural circuits for depression. J Clin Invest. 2009 Apr;119(4):717-25. doi: 10.1172/JCI38454. PMID 19339763
- [Background] Mayberg HS, Brannan SK, Mahurin RK, Jerabek PA, Brickman JS, Tekell JL, Silva JA, McGinnis S, Glass TG, Martin CC, Fox PT. Cingulate function in depression: a potential predictor of treatment response. Neuroreport. 1997 Mar 3;8(4):1057-61. doi: 10.1097/00001756-199703030-00048. PMID 9141092
- [Background] Mayberg HS, Liotti M, Brannan SK, McGinnis S, Mahurin RK, Jerabek PA, Silva JA, Tekell JL, Martin CC, Lancaster JL, Fox PT. Reciprocal limbic-cortical function and negative mood: converging PET findings in depression and normal sadness. Am J Psychiatry. 1999 May;156(5):675-82. doi: 10.1176/ajp.156.5.675. PMID 10327898
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Botteron KN, Raichle ME, Drevets WC, Heath AC, Todd RD. Volumetric reduction in left subgenual prefrontal cortex in early onset depression. Biol Psychiatry. 2002 Feb 15;51(4):342-4. doi: 10.1016/s0006-3223(01)01280-x. PMID 11958786
- [Background] Yucel K, McKinnon M, Chahal R, Taylor V, Macdonald K, Joffe R, Macqueen G. Increased subgenual prefrontal cortex size in remitted patients with major depressive disorder. Psychiatry Res. 2009 Jul 15;173(1):71-6. doi: 10.1016/j.pscychresns.2008.07.013. Epub 2009 May 21. PMID 19464154
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, Crowell AL, Garlow SJ, Rajendra JK, McIntyre CC, Gross RE, Mayberg HS. A connectomic approach for subcallosal cingulate deep brain stimulation surgery: prospective targeting in treatment-resistant depression. Mol Psychiatry. 2018 Apr;23(4):843-849. doi: 10.1038/mp.2017.59. Epub 2017 Apr 11. PMID 28397839
- [Background] Yuan D, Zhao Y, Banks WA, Bullock KM, Haney M, Batrakova E, Kabanov AV. Macrophage exosomes as natural nanocarriers for protein delivery to inflamed brain. Biomaterials. 2017 Oct;142:1-12. doi: 10.1016/j.biomaterials.2017.07.011. Epub 2017 Jul 10. PMID 28715655
- [Background] Boshuizen MCS, Steinberg GK. Stem Cell-Based Immunomodulation After Stroke: Effects on Brain Repair Processes. Stroke. 2018 Jun;49(6):1563-1570. doi: 10.1161/STROKEAHA.117.020465. Epub 2018 May 3. No abstract available. PMID 29724892
- [Background] Detante O, Rome C, Papassin J. How to use stem cells for repair in stroke patients. Rev Neurol (Paris). 2017 Nov;173(9):572-576. doi: 10.1016/j.neurol.2017.09.003. Epub 2017 Oct 21. PMID 29033030
- [Background] Doeppner TR, Bahr M, Hermann DM, Giebel B. Concise Review: Extracellular Vesicles Overcoming Limitations of Cell Therapies in Ischemic Stroke. Stem Cells Transl Med. 2017 Nov;6(11):2044-2052. doi: 10.1002/sctm.17-0081. Epub 2017 Sep 23. PMID 28941317
- [Background] Sarmah D, Agrawal V, Rane P, Bhute S, Watanabe M, Kalia K, Ghosh Z, Dave KR, Yavagal DR, Bhattacharya P. Mesenchymal Stem Cell Therapy in Ischemic Stroke: A Meta-analysis of Preclinical Studies. Clin Pharmacol Ther. 2018 Jun;103(6):990-998. doi: 10.1002/cpt.927. Epub 2017 Dec 14. PMID 29090465
- [Background] Stonesifer C, Corey S, Ghanekar S, Diamandis Z, Acosta SA, Borlongan CV. Stem cell therapy for abrogating stroke-induced neuroinflammation and relevant secondary cell death mechanisms. Prog Neurobiol. 2017 Nov;158:94-131. doi: 10.1016/j.pneurobio.2017.07.004. Epub 2017 Jul 23. PMID 28743464
- [Background] Sussman ES, Steinberg GK. A Focused Review of Clinical and Preclinical Studies of Cell-Based Therapies in Stroke. Neurosurgery. 2017 Sep 1;64(CN_suppl_1):92-96. doi: 10.1093/neuros/nyx329. No abstract available. PMID 28899062
- [Background] Suzuki E, Fujita D, Takahashi M, Oba S, Nishimatsu H. Therapeutic Effects of Mesenchymal Stem Cell-Derived Exosomes in Cardiovascular Disease. Adv Exp Med Biol. 2017;998:179-185. doi: 10.1007/978-981-10-4397-0_12. PMID 28936740
- [Background] Toyoshima A, Yasuhara T, Date I. Mesenchymal Stem Cell Therapy for Ischemic Stroke. Acta Med Okayama. 2017 Aug;71(4):263-268. doi: 10.18926/AMO/55302. PMID 28824181
- [Background] Mah L, Szabuniewicz C, Fiocco AJ. Can anxiety damage the brain? Curr Opin Psychiatry. 2016 Jan;29(1):56-63. doi: 10.1097/YCO.0000000000000223. PMID 26651008
- [Background] McDannold N, Vykhodtseva N, Hynynen K. Blood-brain barrier disruption induced by focused ultrasound and circulating preformed microbubbles appears to be characterized by the mechanical index. Ultrasound Med Biol. 2008 May;34(5):834-40. doi: 10.1016/j.ultrasmedbio.2007.10.016. Epub 2008 Jan 22. PMID 18207311
- [Derived] Mahdavi KD, Jordan SE, Jordan KG, Rindner ES, Haroon JM, Habelhah B, Becerra SA, Surya JR, Venkatraman V, Zielinski MA, Spivak NM, Bystritsky A, Kuhn TP. A pilot study of low-intensity focused ultrasound for treatment-resistant generalized anxiety disorder. J Psychiatr Res. 2023 Dec;168:125-132. doi: 10.1016/j.jpsychires.2023.10.039. Epub 2023 Oct 19. PMID 39491902